CLINICAL TRIAL: NCT03932552
Title: Effects of a Physical Exercise Program on Cerebral and Hepatic Hemodynamics in Patients With Cirrhosis. (Pilot Study)
Brief Title: Effects of a Novel Physical Exercise Program in Patients With Cirrhosis (the LFN-exercise Protocol)
Acronym: LFN-EP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICTLAN-EXERCISE 1
Record Dates: First submitted 2019-03-12; First posted 2019-04-30 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2019-03

CONDITIONS: Cirrhosis; Portal Hypertension; Exercise
MeSH Terms: conditions — Fibrosis; Hypertension, Portal; Motor Activity | interventions — Exercise; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Personalized nutritional therapy
  Interventions: Other: nutritional therapy
- Exercise (Experimental): Aerobic exercise + Personalized nutritional therapy
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — aerobic exercise program during 2 + 12 weeks, highly monitored and tailored to individual physical capacity.
  Arms: Exercise
Other: nutritional therapy — individualised nutritional intervention
  Arms: Control

SUMMARY:
This study evaluates the effects of a structured exercise (The LFN-exercise protocol) program plus diet, on cerebral hemodynamics (cerebral blood flow) and hepatic hemodynamics (portal pressure), as well as on nutritional status (body composition and nutritional markers) in order to facilitate the prescription of exercise in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis of any aetiology (liver biopsy or a combination of clinical and biochemical variables plus evidence of portal hypertension); without decompensation during the past month; serum creatinine <1.5 mg/dL; able to attend the appointed visits and willing to participate in the study.

Exclusion Criteria:

* Presence of high-risk varices in upper endoscopy (red marks, large varices or gastric varices); concomitant cardiopulmonary diseases; decompensated Type 2 Diabetes Mellitus, insulin use or proliferative diabetic retinopathy; orthopaedic or osteomuscular limitations; any type of cancer, primary sclerosing cholangitis and Inflammatory bowel disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Cerebral hemodynamics | 12 weeks
  improvement in transcranial Doppler ultrasound
Improvement in neurocognitive status-1 | 12 weeks
  improvement in neuropsychometric tests (PHES; psychometric Hepatic encephalopathy score)
Improvement in neurocognitive status-2 | 12 weeks
  improvement in neuropsychometric tests (CFF; critical flicker frequency)
Changes in hepatic hemodynamics | 12 weeks
  Improvement in HVPG (HVPG; hepatic venous pressure gradient)
Improvement in body composition | 12 weeks
  improvement in body composition (BIA; Bioelectrical impedance analysis)
Improvement in nutritional status | 12 weeks
  improvement in blood markers of nutritional status (measured in serum/RNA expression)

SECONDARY OUTCOMES:
Physical fitness | 12 weeks
  improvement in 6MWT (6MWT; Six-minute walk test)
Physical activity | 12 weeks
  improvement in Physical activity Questionnaires
Physical activity tolerance | 12 weeks
  improvement in CPET (CPET; Cardiopulmonary exercise test)
Oxidative stress | 12 weeks
  improvement in markers of systemic oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo U Macías-Rodríguez, M.D., PhD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macias-Rodriguez RU, Ruiz-Margain A, Roman-Calleja B, Cantu-Brito C, Flores-Silva F, Gabutti-Thomas A, Aguilar-Najera O, Cruz-Contreras M, Weber-Sangri L, Rios-Torres S, Delgadillo AT, Aguilar-Salinas CA, Kershenobich-Stalnikowitz D. Effect of a monitored exercise protocol in cerebral and hepatic hemodynamics in patients with cirrhosis and portal hypertension. Dig Liver Dis. 2024 May;56(5):827-835. doi: 10.1016/j.dld.2023.11.011. Epub 2023 Nov 25. PMID 38008698